CLINICAL TRIAL: NCT06639230
Title: A Comparative Randomized Clinical Study on the Recurrence Rate of Gingival Pyogenic Granuloma Treated with Sclerotherapy Versus Diode Laser Therapy.
Brief Title: Effect of Laser and Sclerotic Agent in the Treatment of Oral Granuloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nashwa Helaly Mohamed, lecturer, Oral medicine, Periodontology and Oral diagnosis, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oral recurrent granuloma
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pyogenic Granuloma of Gingiva
Keywords: pyogenic granuloma; laser therapy; sclerosing agent
MeSH Terms: conditions — Granuloma, Pyogenic | interventions — Laser Therapy; Sclerotherapy

STUDY DESIGN:
Intervention Model Description: * group 1: This group was made up of ten patients treated using diode lasers with an output power of 3 W in the contact mode, the tip will be moved around the base of the lesion in circles. The base of the lesion was cut precisely till the whole mass was entirely excised.
  * group 2: This group was made up of ten patients who were treated with sclerosing agent after anaesthetizing the surgical site with a local anesthetic agent, the lesion will be injected with the sclerosing agent, diluted in distilled water, the solution is injected slowly into the lesion using a 23-gauge needle until it leaks out from the surface.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Laser-treated group (Active Comparator): 10 patients will be treated by laser surgery to remove oral granuloma
  Interventions: Device: laser therapy
- Sclerotherapy-treated group (group 2) (Active Comparator): This group was made up of ten patients who were treated with injections of sclerosing agent to remove pyogenic granuloma
  Interventions: Drug: Sclerotherapy

INTERVENTIONS:
Device: laser therapy — Laser-treated group (test group): This group consisted of ten patients treated using diode lasers. The diode laser was operated in continuous wave mode with an output power of 3 W in contact mode to excise the pyogenic granuloma. The tip was moved around the base of the lesion in circles. The base of the lesion was cut precisely till the whole mass was entirely excised.
  Arms: Group 1: Laser-treated group
Drug: Sclerotherapy — Sclerotherapy-treated group (control group): This group consisted of ten patients treated with injections of sclerosing agent. After anaesthetizing the surgical site with a local anesthetic agent, The lesion was injected with a 2.5% concentration until it leaked out from the surface, leading to necrosis and spontaneous detachment of the lesion.
  Arms: Sclerotherapy-treated group (group 2)

SUMMARY:
Pyogenic granuloma is a common tumor-like growth of the oral cavity considered to be non-neoplastic in nature. They usually present as a reactive lesion occur in response to chronic and recurring tissue injury, in which capillaries are very prominent commonly seen arising from interdental gingiva. Pyogenic granuloma may occur in all ages, with a peak age of incidence in the second decade of life, more common in young adult females, possibly because of vascular effects of female hormones.

DETAILED DESCRIPTION:
Oral PG can be treated by conservative excision. Local irritants or the source of trauma must be eliminated to minimize the risk of recurrence. Although, surgical excision is considered a simple procedure, it might be complicated by several complications such as intraoperative bleeding, and postoperative infection that might delay the healing of the wound. Other treatment modalities such as laser, injection of sclerosing agents have been used.

Laser has proven to be an effective therapy for oral soft tissue pathologies. Moreover, its ability to perform precise incisions, better hemostasias, and less invasive procedures with less discomfort to patients have made it a preferred treatment option for several soft tissue lesions.

Sclerotherapy has been proposed as an effective method of treatment for pyogenic granuloma. Their mechanism of action is endothelial injury, inflammation, thrombosis, fibrosis, and final lesion destruction. Polidocanol is a widely used nonionic detergent sclerosant that was first developed as an anesthetic. It acts through endothelial overhydration, vascular injury, and closure.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects were principally diagnosed based on history and clinical features such as oral pyogenic granuloma are selected for this study. Radiographic evaluation was also done to rule out any bony involvement.
* The sizes of participants' lesions were not less than 5 mm. • Age > 18 years

Exclusion Criteria:

* Patients were excluded if they had uncontrolled diabetes, renal diseases, coagulation disorders or were allergic to any of the sclerosing drug constituents. Immune-compromised patients and pregnant and lactating women were also excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain was evaluated (NRS) | 3 months
  Postoperative pain intensity will be perceived on the 2nd and 7th days using the ten-point Numeric Rating Scale (NRS) interpreted as 0 grade (No pain), 1-3 grade (mild pain), 4-6 grade (moderate pain) and 7-10 grade (severe pain)
Recurrence rate | 3 months
  Patients will be recalled monthly for 3 months after the end of treatment to evaluate if recurrent occur or not.
Patient compliance (VAS). | 3 months
  compliance of patients will be assessed on a scale from 1 to 10

SECONDARY OUTCOMES:
Details of side effects | 1 week
  details of any side effect as bleeding, oedema, necrosis, infection after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mortada Fikry, professor, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Percutaneous sclerotherapy for vascular malformations: a systematic review — https://pubmed.ncbi.nlm.nih.gov/24509373/
- See also: treatment of intraoral pyogenic granuloma with diode laser 810-980 nm. — https://www.jrmds.in/articles/treatment-of-pyogenic-granuloma-with-diode-laser-91896.html
- See also: Oral pyogenic granuloma: Various concepts of etiopathogenesis. — https://pubmed.ncbi.nlm.nih.gov/22434943/
- See also: Oral Pyogenic Granuloma with Sodium Tetra Decyl Sulphate: A Case Series. — https://pubmed.ncbi.nlm.nih.gov/24027901/